CLINICAL TRIAL: NCT05514964
Title: An Online Intervention to Increase the Ability of LGBT People to Cope With Adverse Events: A Feasibility Study
Brief Title: Interned-delivered Intervention Based on Acceptance Principles
Acronym: LGBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West University of Timisoara (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RO-NO-2019-0412
Record Dates: First submitted 2022-08-22; First posted 2022-08-25 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2022-11

CONDITIONS: Anxiety Disorders; Depression; Mental Health Issue; Well-Being
Keywords: LGBT; online psychological intervention; emotional difficulties; risk factors for anxiety and depression
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Feasibility Studies

STUDY DESIGN:
Intervention Model Description: Feasibility study:
  * An online psychological intervention program (six weeks);
  * Measurement points: Pre-Intervention and Post-Intervention;
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): The experimental arm were provided an intervention program based on John Forsyth & Georg Eifert (2016) The Mindfulness & Acceptance Workbook for Anxiety: A Guide to Breaking Free from Anxiety, Phobias & Worry Using Acceptance & Commitment Therapy, New Harbinger Publications. However, the initial treatment was adapted for the LGBT community using the suggestions from APA Guidelines for Psychological Practice With Lesbian, Gay and Bisexual Clients (2012) and Pachankis, J. E. (2014). Uncovering Clinical Principles and Techniques to Address Minority Stress, Mental Health, and Related Health Risks Among Gay and Bisexual Men. Clinical Psychology: Science and Practice, 21(4), 313-330. doi:10.1111/cpsp.12078.
  Interventions: Behavioral: Feasibility study

INTERVENTIONS:
Behavioral: Feasibility study — Individuals interested to participate in this study were informed about the intervention via the project website and Facebook page of the project. Prior to the start of the study, participants were invited to read the Informed Consent and express their agreement to participate. Only after the Informed Consent was electronically signed, participants were able to complete the screening questionnaires online.
  The intervention program (based on Acceptance and Commitment Therapy) consists of six treatment modules adapted to the online environment. Each module was structured like a therapy session and contained at least two or three homework assignments. Each participant was assigned to an online psychotherapist. At the end of the six modules, participants completed the post-intervention measures.

SUMMARY:
The main objectives for the online intervention were the following:

Designing and implementing an internet-delivered prevention program based on acceptance principles, to support LGBT participants to tackle emotional difficulties more effectively and to become more resilient;

Helping LGBT individuals to remain out of the clinical level of depression and anxiety;

Creating this primary prevention program as a suitable strategy for LGBT individuals to confront emotional difficulties by targeting key risk factors before they evolve further.

DETAILED DESCRIPTION:
This study is part of a research project which addresses a topic under the thematic area of "social sciences and humanities, including gender studies and social inclusion studies." The study targets a particularly disadvantaged group known as the LGBT (lesbian, gay, bisexual, and transgender) community.

The psycho-social and socioeconomic status, in a broader sense, encompasses more than just financial, educational, and occupational aspects. This status also includes the quality of life, an attribute that is consistently dependent on physical and psychological health.

Evidence suggests that people who identify as LGBT are susceptible to various inequalities, including differences in incomes, workplace, and social discrimination. The participants also may suffer from marginalization, poorer mental and physical health, and even legal discrimination (e.g., no recognition of same-sex unions).

This study aims at implementing evidence-based interventions meant to improve the quality of life within the LGBT community. The investigators will also provide mental health support for young LGBT people to cope with potential adverse events.

The implementation of the study will contribute in achieving the three objectives presented above. For instance, by developing and validating an online intervention meant to increase the identity self-acceptance among LGBT participants, the investigators will provide an easily accessible tool to apply the research results with expected positive mental health outcomes for this target group.

ELIGIBILITY:
Inclusion Criteria:

* be fluent in Romanian,
* be at least 18 years of age,
* sexual orientation: gay or bisexual,
* having low or moderate symptoms for at least one of the following self-report scales: generalized anxiety - GAD7 between 5 - 14; social anxiety - SPIN between 21 - 40; depression - PHQ9 between 5 and 14; alcohol - AUDIT between 8 and 14

Exclusion Criteria:

* suicidal ideation (i.e., if exceed a score of 1 on suicide item 9 from PHQ9);
* changes in the dosage if psychotropic medication during the last month (if present),
* have bipolar disorder or psychosis (according to medication status),
* have an alcohol/substance abuse and/or dependence (i.e., AUDIT score > 15),
* have high/clinical levels of anxiety, social anxiety or depression (above the cut-off range - see above)
* currently take part in other psychological treatment,
* obvious obstacle to participation (i.e., no current Internet access, long travel plans during the treatment period etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder-7 (GAD-7) | Change from Pre- to Post-Intervention (6 weeks)
  Generalized Anxiety Disorder 7 (GAD7) was designed to measure participant's level of generalized anxiety or worry. The scale is unidimensional and the total score ranges from 0 to 21. Low scores are associated with low levels of worry, while high scores are associated with high levels of worry.
Social Phobia Inventory (SPIN) | Change from Pre- to Post-Intervention (6 weeks)
  The SPIN scale was designed to measure participant's level of social phobia. The scale is unidimensional and the total score ranges from 0 to 68. Low scores are associated with low levels of social phobia, while high scores are associated with high levels of social phobia.
Patient Health Questionnaire-9 (PHQ-9) | Change from Pre- to Post-Intervention (6 weeks)
  The Patient Health Questionnaire 9 (PHQ9) was designed to measure participant's level of depression. The scale is unidimensional and the total score ranges from 0 to 27. Low scores are associated with low levels of depression, while high scores are associated with high levels of depression.
The Alcohol Use Disorders Identification Test (AUDIT) | Change from Pre- to Post-Intervention (6 weeks)
  The AUDIT scale has 10 questions. Possible responses to each question are scored 0, 1, 2, 3 or 4, with the exception of questions 9 and 10 which have responses of 0, 2 and 4. The range of possible scores is from 0 to 40 where 0 indicates an abstainer who has never had any problems from alcohol. A score of 1 to 7 suggests low risk consumption according to World Health Organization (WHO) guidelines. Scores from 8 to 14 suggest hazardous or harmful alcohol consumption and a score of 15 or more indicates the likelihood of alcohol dependence (moderate-severe alcohol use disorder).

SECONDARY OUTCOMES:
Acceptance and Action Questionnaire 2 (AAQ2) | Change from Pre- to Post-Intervention (6 weeks)
  The AAQ2 scale has 10 items and was designed to measure the ACT's model of mental health and behavioral effectiveness. Scores range from 7 to 49 points, with high scores indicating greater experiential avoidance and immobility.
Brief Multidimensional Experiential Avoidance Questionnaire (BMEAQ) | Change from Pre- to Post-Intervention (6 weeks)
  The 15 items BMEAQ scale was developed to measure the tendency to avoid negative internal experiences. Scores range from 15 to 90 points, with high scores indicating greater tendency in experiential avoidance of the negative feelings.
PTSD Checklist for DSM-5 (PCL-5) | Change from Pre- to Post-Intervention (6 weeks)
  The PCL-5 scale was designed to measure participant's level of post-traumatic stress. The scale is unidimensional and the total score rages from 0 to 80. Low scores are associated with low levels of post-traumatic stress, while high scores are associated with high levels of post-traumatic stress.
Internalized Homophobia Scale (IHS) | Pre-Intervention
  The Internalized Homophobia Scale has 26 items and was designed to measure the internalized homonegativity. The items are scored on a Likert-type scale from 0 "strongly disagree" to 6 "strongly agree". The total score rages from 0 to 156, where high scores are associated with high levels of internalized homophobia.
Sexual Orientation Concealment Scale (SOCS6) | Pre-Intervention
  The Sexual Orientation Concealment Scale is a 6 items measure designed to assess lesbian, gay and bisexual (LGB) individual's active concealment of their sexual minority status. Averaging the six items produces the overall SOCS score, which ranges from 0 to 24, where high scores are associated with high levels of concealment.
Daily Heterosexist Experiences Questionnaire (DHEQ) | Pre-Intervention
  The Daily Heterosexist Experiences Questionnaire has 50 items and they are scored on a Likert-type scale from 0 "It didn't happen to me/It doesn't apply to me" to 5 "It happened to me and it bothered me a lot". The measure can be scored in two ways:
  1. Occurrence: Responses are recoded 0 = 0 (did not occur) and 1 through 5 = 1 (did occur). Items are then summed for a total score indicating how many of these experiences participants have had.
  2. Distress: Responses are recoded so that 0 and 1 = 1 (did not bother) and the rest of the responses remain the same. A mean is then computed for responses to all items, indicating the mean level of distress participant feels related to these experiences.
  The scale has nine subscales: Vigilance, Harassment and discrimination, Gender expression, Parenting, Victimization, Family of origin, Vicarious trauma, Isolation and HIV/AIDS.

CONTACTS AND LOCATIONS:
Locations (1):
- West University of Timisoara, Timișoara, Romania

REFERENCES:
- [Derived] Isbasoiu AB, Sava FA, Larsen TMB, Anderssen N, Rotaru TS, Rusu A, Salagean N, Tulbure BT. An Internet-Based Intervention to Increase the Ability of Lesbian, Gay, and Bisexual People to Cope With Adverse Events: Single-Group Feasibility Study. JMIR Form Res. 2024 May 15;8:e56198. doi: 10.2196/56198. PMID 38749024
- See also: The Romanian website where the program was implemented. — https://www.e-cbt.ro/program/PACT/programul-pact